CLINICAL TRIAL: NCT00984919
Title: Pilot Study of the Role of 11-dh-TXB2 in Prostate Cancer Screening and Diagnosis
Brief Title: Biomarker 11-dh-TXB2 in Blood and Urine Samples From Patients With Prostate Cancer and Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Elisabeth Heath, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Other Study IDs: CDR0000654093; P30CA022453 (NIH); WSU-2009-058
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer; stage I prostate cancer; stage II prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Chromatography, High Pressure Liquid; Mass Spectrometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: high performance liquid chromatography
Other: laboratory biomarker analysis
Other: mass spectrometry

SUMMARY:
RATIONALE: Studying samples of blood and urine from patients with cancer in the laboratory may help doctors identify biomarkers related to cancer.

PURPOSE: This research study is looking at a biomarker, 11-dh-TXB2, in blood and urine samples from patients with prostate cancer and healthy volunteers.

DETAILED DESCRIPTION:
OBJECTIVES:

* To identify a potential novel marker of prostate cancer in the blood and urine, 11-dh-TXB2, to be used as a screening tool for prostate cancer as well as in detection of early relapse in patients previously treated for early-stage prostate cancer.

OUTLINE: Blood and urine samples are collected and analyzed for plasma and urinary 11-dh-TXB2 levels by HPLC and tandem-mass spectrometry.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets one of the following criteria:

  * Histopathologically confirmed prostate cancer meeting 1 of the following criteria:

    * Newly diagnosed untreated disease
    * Received prior local therapy (prostatectomy, definitive radiotherapy, brachytherapy, or cryotherapy) with no evidence of disease activity (defined as serum PSA < 0.4 ng/mL post therapy) and by imaging studies
    * Experienced biochemical failure (defined as rise in serum PSA ≥ 0.4 ng/mL post therapy)
  * Healthy volunteer (clinic patient with no history of clinically significant malignancies within the past 6 months)

PATIENT CHARACTERISTICS:

* No clinical evidence of liver cirrhosis or chronic liver disease (i.e., evidence of ascites or severe coagulopathy)
* No active prostatitis

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 30 days since prior and no concurrent regular antiplatelet agents (including aspirin, anagrelide, cilastazole, clopidogrel, dipyridamole, pentoxiphylline, sulfinpyrazone, or ticlopidine)
* More than 7 days since prior and no concurrent NSAIDs (including ibuprofen, celecoxib, diclofenac, diflunisal, etodolac, fenoprofen, flurbiprofen, indomethacin, ketoprofen, meclofenamate, mefenamic acid, nabumetone, naproxen, oxaprozin, piroxicam, sulindac, or tolmetin)

Ages: 40 Years to 120 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cancer clinic
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-11; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Identification of 11-dh-TXB2 in the blood and urine | 2 to 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth I. Heath, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States